CLINICAL TRIAL: NCT04586257
Title: Effect of Thoracolumbar Interfacial Plane Block or Erector Spinae Plane Block on the Enhanced Recovery After Spine Surgeries: Prospective Randomized Double-blind Study
Brief Title: Effect of Regional Anesthesia on Enhanced Recovery After Spine Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 34142/9/20
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: ERAS
Keywords: Spine surgery; Length of hospital stay; ERAS; Regional analgesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * The patients will be blinded to their groups.
  * An anesthesia resident who will not participate in the study and have no subsequent rule in it will help in the preparation of local anesthetic mixtures under strict aseptic precautions.
  * An assistant nurse who will be blinded to the study groups and will have no subsequent rule in it will help in the collection of the data of measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): patients in this group will receive Erector spinae plane block after induction of general anesthesia.
  Interventions: Procedure: Erector spinae plane block
- Group II (Experimental): patients in this group will receive thoracolumbar interfascial plane block after induction of general anesthesia
  Interventions: Procedure: Throacolumbar interfacial plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — While patients in the prone position, 1.4-5.1 MHz low-frequency probe (C5-1s convex transducer) will be first placed in a longitudinal orientation in the midline to identify the spinous process of at the appropriate lumbar level, then it will be scanned laterally about 2-3 cm until visualization of the paraspinal muscles and the transverse process at the same time. After standard sterilization, a 21-G short bevel nerve block needle will be advanced in a cephalad-to-caudal direction, in-plane under real- time ultrasound guidance, through skin, subcutaneous tissue, and erector spinae muscles until reaching the transverse process. After negative aspiration of blood or cerebral spinal fluid, a small volume of local anesthetic was injected to confirm the position of the needle tip between the erector spinae muscles and the transverse process. A total of 20 ml of 0.0.25% plain bupivacaine will be incrementally injected with intermittent negative aspiration on each side.
  Arms: Group I
Procedure: Throacolumbar interfacial plane block — USG-guided TLIP block will be performed using a high-frequency linear probe while the patient in prone position. The probe will be covered with sterile sheath positioned transversally in a midline position at approximately the level of the 3rd lumbar vertebra (L3). The corresponding spinous process and interspinal muscles will be identified, and the probe will be slid laterally to identify the multifidus (MF) muscle and longissimus (LG) muscle. Sliding the probe from midline to laterally helps in the correct identification of various muscles. After identifying the muscles, TLIP block will be performed aseptically on both sides of L3 vertebra. Under ultrasound guidance, an insulated echogenic needle will be inserted in-plane in a lateral to medial orientation in-plane USG guided through the belly of LG toward the MF. When needle reach deep to middle of MF/LG interface, 20 ml 0.25% bupivacaine will be injected after negative aspiration. The block will be administered bilaterally.
  Arms: Group II

SUMMARY:
This study will be carried out on 80 patients who will be presented for different spine surgeries under general anesthesia and regional anesthesia technique in Tanta university hospitals. The study was approved by the research ethics committee of the faculty of medicine.

Patients will be admitted to the OR where induction of general anesthesia was started and then, the patients will be randomly distributed into two equal groups; -

* Group I (40 patients) (ESP block): patients in this group will receive ESP block after induction of general anesthesia.
* Group II (40 patients) (TLIP block): patients in this group will receive TLIP block after induction of general anesthesia

Measurements; - The length of hospital stay as the primary outcome Postoperative pain scores and opioid consumption as the Secondary outcome

DETAILED DESCRIPTION:
This prospective randomized double-blind study will be carried out on 80 adult patients who will be presented for different spine surgeries in Tanta university hospitals after obtaining the approval from the institutional Ethical Committee, informed written consent will be obtained from all the participants.

Patients will be randomly classified using a computer-generated software of randomization into 2 groups:

* Group I (40 patients) (ESP block): patients in this group will receive ESP block after induction of general anesthesia.
* Group II (40 patients) (TLIP block): patients in this group will receive TLIP block after induction of general anesthesia

Anesthetic technique

* The patients will be assessed preoperatively in the anesthesia clinic. On arrival of patients to the preparation room, an intravenous line will be established and the patient will be connected to a monitor. All the patients will receive pheniramine hydrogen maleate 45.5 mg intravenous as an antihistamine, Cefazolin30 mg/kg, and 40 mg pantoprazole.
* Induction of anesthesia will be carried out by fentanyl 1 ug/kg, propofol 1.5 mg/kg, and atracurium 0.5 mg/kg to facilitate tracheal intubation. After securing the airway through a suitable sized endotracheal tube, the patient was connected to a mechanical ventilator with its parameters adjusted to maintain the end-tidal carbon dioxide 34-38 mmHg.
* Maintenance of the anesthesia was performed by isoflurane 1.MAC and incremental doses of atracurium 0.1 mg/kg. A temperature probe was inserted in the nasopharynx for core temperature monitoring. The depth of anesthesia was monitored by the bispectral index (Covidien, Mansfield, MA, USA). The BIS values were kept 40-60. An additional bolus dose of fentanyl 0.5 ug/kg was used in case of increase BIS more than 60 or increase in the heart rate or mean arterial pressure by more than 15 % of the baseline values.
* All patients received tranexamic acid 30 mg/kg through intravenous infusion. Before skin incision, patients of group I will receive ultrasound-guided ESP block, while patients in group II will receive ultrasound guided TLIP block.
* At the end of the surgery, the isoflurane was switched off with reversal of muscle relaxation and awake tracheal extubation and transfer of the patient to the recovery room for postoperative monitoring and supplementation of oxygen through a nasal cannula (2-3 L/min). All the patients will receive 4 mg dexamethasone I .v after induction of anesthesia and 4 mg of ondansetron i.v at the end of the surgery to guard against postoperative nausea and vomiting. All the patients received routine postoperative analgesia in the form of paracetamol 1 gm i.v infusion every 6 hours and ketorolac 30 mg i.v every 12 hours. Rescue analgesia in the form of morphine 3 mg i.v was administrated when the pain score was more than 3.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes aged (21-70 years) with ASA physical status I-III scheduled for spine surgeries.

Exclusion Criteria:

* Patient refusal
* Body mass index (BMI) less than 18 or higher than35 kg/m2
* Pregnant
* History of relevant allergy to related perioperative medications
* Previous lumbar spine surgery
* Existing contraindications to nerve block such as coagulopathy, local and systemic infection
* Hepatic or renal insufficiency
* Chronic opioid use

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | Within 7 days of the surgery
  The time interval in days from the day of the surgery till discharge of the patient from the hospital.

SECONDARY OUTCOMES:
postoperative pain scores | Within the first 24 hours after surgery
  Postoperative Numerical rating score (NRS) every 2 hours in the first six hours, then every 4 h till 24 h. When NRS scores reach 4 or more, 3 mg of i.v morphine will be given and can be repeated if required with calculation of the total postoperative morphine consumption in mg in the first 24 hours after surgery and the time to the first request of rescue analgesia
The postoperative opioid consumption | Within the first 24 hours after surgery
  The total dose of morphine consumed in the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Abdelkhalik, Principal Investigator — Tanta University
Locations (1):
- Faculty of Medicine, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data of primary outcome will be available with the corresponding author till 6 months after approval of the publication of the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data of primary outcome will be available with the corresponding author till 6 months after approval of the publication of the trial.
Access Criteria: Contact the principal investigator